CLINICAL TRIAL: NCT06697353
Title: ROVER Japan/ Real-world Outcomes of Patients Treated With Vericiguat in Japanese Routine Care: a Retrospective Cohort Study Using a Hospital Administrative Database
Brief Title: An Observational Study to Learn More About the Real-world Outcomes in Patients With Heart Failure Who Initiate Treatment With Vericiguat in Japan
Acronym: ROVER Japan
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22849
Record Dates: First submitted 2024-10-31; First posted 2024-11-20 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Chronic Heart Failure; Chronic Heart Failure With Reduced Ejection Fraction
Keywords: HFrEF
MeSH Terms: interventions — vericiguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (15):
- Study Cohort: Patients who initiated on-label use of vericiguat (i.e. patients treated with at least one HF therapy who initiated vericiguat with a starting dose of 2.5 mg). Adult patients with Heart Failure (HF) diagnosis code between March 2021 and July 2024, initiating vericiguat between September 2021 and July 2024, with HF diagnosis prior to index date, and with at least 180 days of observation prior to index date.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort a: derived from the study cohort, and defined as: With (a1) /without (a2) recent worsening of HF (WHF). With recent WHF will be defined as HF hospitalization within 6 months or outpatient intravenous diuretic dispensation (Anatomical Therapeutic Chemical (Classification System) (ATC) codes C03 and receipt code) within 3 months.
  Without recent WHF will be defined as no HF hospitalization for 6 months and no outpatient Intravenous (IV) diuretic use for 3 months
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort b: derived from the study cohort, and defined as: Time from WHF event to vericiguat initiation. Within patients with recent WHF, patients will further be classified according to the timing from WHF event as: HF hospitalization in the previous 3 months, HF hospitalization in the previous 3-6 months, and outpatient IV diuretics (without HF hospitalization) in the previous 3 months.
  Note that patients who have a record of hospitalization both in the previous 3 months and the previous 3-6 months will be classified in "HF hospitalization in the previous 3-6 months.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort c: derived from the study cohort, and defined as: With (c1)/without (c2) Angiotensin Receptor Neprilysin Inhibitor (ARNI). With ARNI will be defined as presence of prescription or dispensation of sacubitril/valsartan (ATC code C09DX04), within the 90 days prior to index date (exclusive).
  Without ARNI will be defined as absence of prescription or dispensation of sacubitril/valsartan (ATC code C09DX04), within the 90 days prior to index date (exclusive).
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort d: derived from the study cohort, and defined as: With (d1)/without SGLT2i (d2). With SGLT2i will be defined as presence of prescription or dispensation of dapagliflozin (ATC code A10BK01) and empagliflozin (ATC code A10BK03) within the 90 days prior to index date (exclusive).
  Without SGLT2i will be defined as absence of prescription or dispensation of dapagliflozin (ATC code A10BK01) and empagliflozin (ATC code A10BK03) within the 90 days prior to index date (exclusive).
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort e: derived from the study cohort, and defined as: Number of foundational therapies (i.e., ACEi, ARB, ARNI, ACEi/ARB, ACEi/ARB/ARNI, BB, MRA and SGLT2i). Presence/absence of each foundational therapy - ACEi (enalapril [ATC code C09AA02] and lisinopril [ATC code C09AA03]), ARB (candesartan [ATC code C09CA06]), ARNI (sacubitril-valsartan [ATC code C09DX04]), ACEi/ARB, ACEi/ARB/ARNI, BB (bisoprolol [ATC code C07AB07] and carvedilol [ATC code C07AG02]), MRA (spironolactone [ATC code C03DA01] and eplerenone [ATC code C03DA04]) and SGLT2i (dapagliflozin [ATC code A10BK01] and empagliflozin [ATC code A10BK03]) - will be assessed within the 90 days prior to index date (exclusive).
  The number of foundational therapies present will be categorized by none, mono therapy, dual therapy, triple therapy, and quadruple therapy.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort f: derived from the study cohort and defined as: Age group. Age group will be categorized as <65, 65 to <75, and ≥75 years
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort g: derived from the study cohort, and defined as: sex (will be categorized as male and female)
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort h: derived from study cohort and described as: Body mass index categories. Body mass index is defined as a person's weight in kilograms divided by the square of the person's height in meters (kg/m2), and will be categorized as underweight (<18.5 kg/m2), normal weight (18.5-24.9 kg/m2), pre-obesity (25.0-29.9 kg/m2), and obesity (≥30.0 kg/m2).
  The body mass index value closest to the index date and prior to the index date will be used for this classification. If multiple body mass index values exist, the value closest to the index date will be used.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort i: derived from study cohort and described as: With chronic kidney disease (all; stage ≥3). With chronic kidney disease (CKD) will be defined by the presence of the N18 International Classification of Diseases, 10th revision (ICD-10 code( within 180 days prior to index date . A subset of CKD stage ≥3 will be identified with the N18.3-N18.5 ICD-10 codes.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort j: derived from study cohort and described as: Up-titration level of vericiguat at 3 months. Up-titration level for vericiguat at 3 months of treatment will be categorized as vericiguat dosage: 2.5 mg, 5 mg, 10 mg or other dose.
  Note that when patients' up-titration level has increased to the upper level within 3 months, unless the level at 3 month remains at the upper level, the patients will not be considered up-titrated.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort k: derived from study cohort and described as: Adherent (k1) vs. non-adherent (k2) to vericiguat within 3 months. Adherence to vericiguat within 3 months of treatment will be defined as a medication possession ratio (MPR) of ≥80%.
  Non-adherent to vericiguat within 3 months of treatment will be defined as MPR<80% .
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub-Cohort l: derived from study cohort and described as: Persistent (l1) vs. non-persistent (l2) to vericiguat within 3 months. Treatment discontinuation within 3 months of treatment will be identified by a gap of >30 days between successive prescription records or between the last prescription record and the end of follow-up. Persistent within 3 months will be defined as no treatment discontinuation within 3 months of treatment.
  Non-persistent within 3 months to vericiguat will be defined as treatment discontinuation within 3 months of treatment.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub Cohort m: derived from study cohort and described as: Index date categories. Patients will be classified according to the year of inclusion as follows: September 2021 to August 2022 vs. September 2022 to July 2024.
  Interventions: Drug: vericiguat (BAY 1021189)
- Sub Cohort n: derived from the study cohort and described as: Discontinuing ARNI before initiating vericiguat. Patients with a prescription/dispensation of ARNI within the 90 days prior to index date (exclusive) and no prescription/dispensation of ARNI within the 90 days after the index date (inclusive).
  Interventions: Drug: vericiguat (BAY 1021189)

INTERVENTIONS:
Drug: vericiguat (BAY 1021189) — 2.5 mg initiating dose
  Other Names: VERQUVO

SUMMARY:
This is an observational study in which data already collected from people with chronic heart failure is studied.

Chronic HFrEF is a long-term condition where the left side of the heart does not pump blood out to the body as well as it should. Blood and fluid may collect in the lungs, blood vessels, and tissues causing shortness of breath or tiredness. Over time, heart failure can lead to other serious medical conditions that may result in hospital stays or even death.

The study drug, vericiguat, is already approved for doctors to prescribe to people with chronic HFrEF in Japan.

Vericiguat increases the activity of an enzyme called soluble guanylate cyclase (sGC), which relaxes the blood vessels, allowing more blood to flow through. As a result, the heart is able to pump better.

The participants in this study are already receiving treatment with vericiguat (newly initiated) as part of their regular care from their doctors.

There is currently limited real-world data on the use of vericiguat in Japanese people. Therefore, more research is needed on larger groups of Japanese people for a longer period to understand the effects of use of vericiguat.

The main purpose of this study is to collect information about how well vericiguat is used in Japanese people with heart failure who initiate vericiguat treatment.

To do this, researchers will collect the following information for participants who newly initiated vericiguat:

occurrence of death due to heart and blood vessel related events

occurrence of death due to any reason

hospital stays due to heart failure

a combination of hospital stays due to heart failure or occurrence of death due to heart and blood-vessel related events

a combination of occurrence of death due to any reason or hospital stays due to heart failure

In addition, researchers will collect the following information:

participants' characteristics, including age, sex, height, weight, and medical history

how well did the participants follow their prescribed treatment with vericiguat over the year after starting it

how long did the participants continue to take vericiguat over the year after starting it

changes in the dose of vericiguat in the participants over the year after starting it

other treatment options participants have taken for the treatment of heart failure

changes in laboratory values and other test results before and after treatment with vericiguat

The data will come from the participants' hospital records provided by the Medical Data Vision Co., Ltd. They will cover the period from September 2016 to July 2024.

Researchers will track participants' data and will follow them for a maximum of one year after starting treatment with vericiguat, or until any of the following happens:

the participant dies

the participant cannot be tracked anymore

the end of the study

In this study, only available data from routine care are collected. No visits or tests are required as part of this study.

ELIGIBILITY:
Inclusion Criteria:

Patients who initiate vericiguat (identified by Anatomical Therapeutic Chemical [ATC] code C01DX22, generic name and receipt code [to be defined in the SAP]) between September 2021 and July 2024

* Patients who have diagnosis code of HF (identified by World Health Organization [WHO] International Classification of Diseases, 10th revision [ICD-10] codes I50, I11.0) prior to index date
* Patients aged 18 years or older at index date

Exclusion Criteria:

* Patients with observability for less than 180 days prior to index date
* Patients with a follow-up period of 0 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population is composed of adult patients with HF diagnosis code between March 2021 and July 2024, initiating vericiguat between September 2021 and July 2024, with HF diagnosis prior to index date, and with at least 180 days of observation prior to index date.
Sampling Method: Probability Sample
Enrollment: 4936 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-09-19 (Actual); Study Completion 2025-09-19 (Actual)

PRIMARY OUTCOMES:
Incidence rates of clinical outcomes in patients who initiate vericiguat | Retrospective analysis from September 2016 to July 2024; Up to one year after vericiguat initiation
  To estimate the incidence rates of cardiovascular death, all-cause death, HF hospitalization, a composite of cardiovascular death or HF hospitalization, and a composite of all-cause death or HF hospitalization in patients who initiate vericiguat

SECONDARY OUTCOMES:
characteristics of patients who initiate vericiguat: age | Baseline
  Age in years: to document the age range of patients initiating vericiguat
characteristics of patients who initiate vericiguat: gender | Baseline
  Gender: to document the gender distribution of patients initiating vericiguat
characteristics of patients who initiate vericiguat: BMI | Baseline
  BMI (in kg/m2) at baseline - To describe the weight distribution of patients who initiate vericiguat
characteristics of patients who initiate vericiguat: recent Worsening Heart failure (WHF) | Baseline
  Documentation of Recent WHF event: HF hospitalization within 6 months or outpatient IV diuretics within 3 months prior to index date.
characteristics of patients who initiate vericiguat, prior WHF | Baseline
  Prior WHF: HF hospitalization or outpatient IV diuretics with no specified evaluation period
characteristics of patients who initiate vericiguat: Dialysis | Baseline
  Document the number of patients on maintenance dialysis
characteristics of patients who initiate vericiguat: Time from recent WHF event | Baseline
  Treatment location after recent WHF event: HF hospitalization in the previous 3 months, HF hospitalization in the previous 3-6 months, and outpatient IV diuretics in the previous 3 months
characteristics of patients who initiate vericiguat: Comorbidities | Baseline
  Document Comorbidities at baseline
characteristics of patients who initiate vericiguat: setting | Baseline
  Setting of vericiguat initiation: inpatient or outpatient setting - To describe the characteristics of patients who initiate vericiguat
characteristics of patients who initiate vericiguat: cardiovascular procedure | Baseline
  Document Cardiovascular procedures
characteristics of patients who initiate vericiguat: HF foundational therapy, prior index date | Baseline
  HF foundational therapy within 90 days prior to index date
characteristics of patients who initiate vericiguat: Number of HF foundational therapy | Baseline
  Number of HF foundational therapy within 90 days prior to index date
adherence of vericiguat therapy for 1 year after treatment initiation: medication possession ratio (MPR) | 1 year (after vericiguat initiation)
  To describe the adherence of vericiguat therapy for 1 year after treatment initiation measured by medication possession ratio (MPR)
adherence of vericiguat therapy for 1 year after treatment initiation: proportion of days covered (PDC) | 1 year (after vericiguat initiation)
  To describe the adherence of vericiguat therapy for 1 year after treatment initiation measured by proportion of days covered (PDC)
persistence of vericiguat therapy for 1 year after treatment initiation: Duration of continuous treatment over the first year after the index date | 1 year (after vericiguat initiation)
  To describe the persistence of vericiguat therapy for 1 year after treatment initiation measured by the duration of continuous treatment
persistence of vericiguat therapy for 1 year after treatment initiation: percentage of patients with continuous treatment at Day 365 | 1 year (after vericiguat initiation)
  To describe the persistence of vericiguat therapy for 1 year after treatment initiation measured by the percentage of patients with continuous treatment at Day 365
Pattern description of dose titration of vericiguat over 1 year after treatment initiation: Day-to-day patterns of vericiguat | 1 year (after vericiguat initiation)
  To describe the patterns of dose titration of vericiguat over 1 year after treatment initiation measured by day-to-day patterns
Pattern description of dose titration of vericiguat over 1 year after treatment initiation: Time to up-titration of vericiguat from index date to Day 365 | 1 year (after vericiguat initiation)
  To describe the patterns of dose titration of vericiguat over 1 year after treatment initiation measured by time to up-titration
Pattern description of dose titration of vericiguat over 1 year after treatment initiation: Time to up-titration to maximal daily dose of vericiguat from index date to Day 365 | 1 year (after vericiguat initiation)
  To describe the patterns of dose titration of vericiguat over 1 year after treatment initiation measured by time to up-titration to maximal daily dose
Pattern description of Heart Failure (HF) therapy before and after vericiguat initiation | Baseline and 1 year (after vericiguat initiation)
  To describe the patterns of HF therapy before and after vericiguat initiation
Pattern description of dose titration of HF therapy before and after vericiguat initiation | Baseline and 1 year after vericiguat initiation
  To describe the patterns of dose titration of HF therapy before and after vericiguat initiation
assess the change in laboratory and clinical parameters before and after vericiguat initiation | Baseline and 180 days after vericiguat initiation
  To assess the change in laboratory and clinical parameters before and after vericiguat initiation measured by SBP, LVEF, NYHA classification, NT-proBNP, BNP, eGFR, hemoglobin, number of HF hospitalization per patient, dose of diuretics, and number and percentage of patients with diuretic use.

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.

REFERENCES:
- See also: Related Info — https://clinicaltrials.bayer.com/study/22849